CLINICAL TRIAL: NCT07054294
Title: Study on Total Energy Expenditure and Its Influencing Factors in Chinese Children Aged 7-13 Years (Including Rural Areas) Using the Doubly Labelled Water Method
Brief Title: Total Energy Expenditure Across the Life Course in Low-and Middle-Income Countries -- Chinese Children
Status: Recruiting | Type: Observational
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Xueying Zhang, Associate researcher, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Other Study IDs: SIAT-IRB-241115-H0927
Record Dates: First submitted 2025-06-17; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine samples will be collected from children over a 14-day period following the administration of doubly labeled water (DLW). The analysis of oxygen-18 and deuterium in these urine samples will be used to calculate the total energy expenditure of the children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By 2050, there will be 9 billion people on earth. It will be necessary to feed them to avoid the population catastrophe predicted by Malthus 150 years ago. Yet a major issue facing governments is that the current method by which food demands are estimated is widely acknowledged as completely inaccurate. An accurate method is available. It is based on measurements of isotope elimination, called the doubly labelled water (DLW) method. In 2018, the International Atomic Energy Agency (IAEA) hosted and compiled a database of measurements using this technique. It showed that the use of the DLW method has been mostly restricted to the USA and Western Europe. It has rarely been applied across Africa and Asia. The database also focused on adults, leaving much unknown about the energy balance in children and adolescents. There is a clear need to fill this gap in knowledge, providing information that governments across Low- and Middle-Income countries can use to forecast future food demands. In China, the prevalence of overweight and obesity among children and adolescents is increasing. In 2009, 22.1% of Chinese youth aged 7-17 years were either overweight or obese, according to the China Health and Nutrition Survey. The obesity rate has increased fourfold since 1995. One of the most concerning problems is the persistence of childhood obesity into adulthood. The causes of this obesity epidemic are strongly disputed, with some suggesting it is due to increasingly sedentary lifestyles (computers, cars, phones, etc.), while others suggest it is mostly due to changing food patterns (junk food and sugar-sweetened beverages). Measuring energy expenditure in children and adolescents in China will address whether declining expenditure due to reduced physical activity is a key cause of the epidemic. Most measurements come from urban populations, leaving rural populations greatly underrepresented.

DETAILED DESCRIPTION:
The investigators will recruit healthy Chinese children aged 7-13 years to participate in a study investigating growth and energy needs. Each participant will complete basic anthropometric measurements-including height, weight, waist and hip circumference, and mid-upper arm circumference. Questionnaires will be used to assess family socioeconomic status, dietary intake, and pubertal development. The investigators will also measure total energy expenditure, basal metabolic rate, physical activity, body composition, and environmental temperature exposure.

This research will provide accurate data on the energy expenditure of children and adolescents living in China. These data will inform national estimates of food and energy requirements, support public health nutrition strategies, and help fill critical data gaps in the IAEA Doubly Labeled Water (DLW) database.

Study Details Anthropometric Measurements

1. Height: Height will be measured using a Seca 217 stadiometer. Participants will stand barefoot with feet approximately 60° apart. Heels, sacrum, and shoulder blades will be placed against the stadiometer's vertical rod. The head will be aligned so that the upper margin of the ear canal is level with the lower margin of the eye socket. The horizontal plate will be lowered gently to rest on the crown of the head. Two measurements will be taken and averaged; values will be recorded to the nearest 0.1 cm.
2. Body Weight: After an overnight fast, body weight will be measured in the morning using a calibrated TANITA MC-780 scale. Participants will wear light clothing and no shoes.
3. Waist Circumference: Waist circumference will be measured at the midpoint between the iliac crest and the lower edge of the 12th rib. Participants will stand with feet 25-30 cm apart and body weight evenly distributed. A flexible tape will be wrapped snugly (without compression), and two measurements will be averaged to the nearest 0.1 cm.
4. Hip Circumference: Hip circumference will be measured with the participant standing straight, legs together, arms relaxed. The tape will be placed horizontally at the level of the pubic symphysis and the most prominent part of the buttocks. Two measurements will be taken and averaged.
5. Mid-Upper Arm Circumference: The participant will stand or sit upright with the arm relaxed. The midpoint between the acromion (shoulder) and olecranon (elbow) will be marked. A measuring tape will be wrapped around this midpoint with light contact. Two measurements will be taken and averaged.

Questionnaires

1. Family Socioeconomic Status: Will be assessed using a structured SES questionnaire.
2. Pubertal Development: Will be assessed via Tanner staging for secondary sexual characteristics.
3. Dietary Intake: Will be assessed using three 24-hour dietary recall questionnaires administered on non-consecutive days.

Body Composition (BIA) Bioelectrical impedance analysis (TANITA MC-780) will be used to measure segmental weight (arms, legs, trunk), total body fat percentage (fat%), fat mass (FM), fat-free mass (FFM), total body water (TBW), muscle mass, and BMI.

Basal Metabolic Rate Basal metabolic rate (BMR) will be measured using indirect calorimetry via a Cosmed Quark system with a ventilated hood. After a 10-hour overnight fast and no strenuous activity in the preceding day, participants will lie supine under the hood for 30 minutes. Oxygen consumption and carbon dioxide production will be monitored, and the final 10 minutes will be used to calculate BMR (Weir, 1949). Equipment will be validated monthly via alcohol burn tests and turbine flow calibration.

Total Energy Expenditure (DLW Method) Total energy expenditure (TEE) will be measured using the doubly labeled water (DLW) method. Urine samples will be collected and stored at -20 °C, then shipped on dry ice to Dr. John Speakman's laboratory at the University of Aberdeen or to the Shenzhen Institute of Advanced Technology. Isotope ratios will be analyzed using a near-infrared isotope gas analyzer. Mean CO₂ production will be calculated using equations developed by Speakman et al. (2021), and TEE will be derived using the Weir equation (1949).

Environmental Temperature Exposure Environmental exposure will be monitored using iButton sensors (DS1921G). These will be placed in the participant's living environment (e.g., on a backpack, clothing, indoor wall, or building exterior) using waterproof medical-grade adhesive. This will allow measurement of ambient temperature during the study period.

Physical Activity Physical activity will be monitored using ActiGraph GT3X accelerometers worn at the waist for 14 consecutive days, except during water activities (e.g., bathing or swimming). Data will be considered valid if the monitor is worn for at least 12 hours on four days, including at least two weekdays and two weekend days. The first day of wear and any day with insufficient data will be excluded from analysis.

ELIGIBILITY:
Inclusion Criteria:

-Healthy participants

Exclusion Criteria:

1. Malnutrient as defined by the Chinese national standards WS/T 456-2014 and WS/T 586-2018

   1. Nutritional deficiencies
   2. Overweight
   3. Obesity
2. Acute illness within the past 7 days

   1. Fever
   2. Diarrhea
   3. Vomiting
3. Chronic diseases

   1. Cardiovascular diseases
   2. Diabetes mellitus or any form of metabolic disorders

      * Type 1 or Type 2 diabetes
      * Metabolic syndrome
      * Hyperlipidemia
      * Dyslipidemia
   3. Renal diseases

      * Chronic kidney disease
      * Nephrotic syndrome
4. Musculoskeletal injuries
5. Disabilities

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of healthy children aged 7 to 13 years who exhibit normal growth and development. Participants will neither be overweight nor obese, nor will they have any nutritional deficiencies. They will be capable of cooperating to complete all required measurements. None of the children will have been diagnosed with chronic diseases or musculoskeletal injuries or disabilities. Additionally, all participants will be free from acute clinical illnesses for at least seven days prior to the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Height | About 3 minutes.
  Height in centimetres will be measured by Leicester stadiometer(Seca 217, Germany).
Weight | About 5 minutes.
  Weight in kilograms will be measured by TANITA.
BMI | About 10 minutes (calculated).
  BMI values in kg/m2 were calculated from weight measured by TANITA and height measured by Leicester stadiometer (Seca 217, Germany).
Fat mass | About 3 minutes.
  Fat mass in kilograms will be measured by TANITA.
Fat percentage | About 3 minutes.
  Fat percentage will be measured by TANITA.
Fat-free mass | About 3 minutes.
  Fat-free mass in kilograms will be measured by TANITA.
Muscle mass | About 3 minutes.
  Muscle mass in kilograms will be measured by TANITA.
Total body water | About 3 minutes.
  Total body water in kilograms will be measured by TANITA.
Anthropometric measurements | About 10 minutes.
  Anthropometric measurements, including waist circumference (measured in centimeters), will be obtained using a flexible tape measure following standardized protocols.
Anthropometric measurements | About 10 minutes.
  Anthropometric measurements, including hip circumference (measured in centimeters), will be obtained using a flexible tape measure following standardized protocols.
Anthropometric measurements | About 10 minutes.
  Anthropometric measurements, including mid-upper arm circumference (measured in centimeters), will be obtained using a flexible tape measure following standardized protocols.
Family socioeconomic status | About 5 minutes.
  Family socioeconomic status will be assessed by the Family Socioeconomic Status Questionnaire (SES).
Secondary sexual characteristics | About 5 minutes.
  The Tanner stages are used to assess the development of secondary sexual characteristics and are divided into five stages. For boys, the evaluation includes pubic hair development and genital development (including testicular and penile growth). For girls, the evaluation includes pubic hair development and breast development (thelarche).
Dietary intake | About 10 minutes (three times).
  The 24-hour dietary recall questionnaire is used to investigate the dietray intake level of the subjects. Three daily meals will be collected to calculate the dietary intake in kcal or MJ.
Basal metabolic rate | About 30 minutes.
  The basal metabolic rate in kcal or MJ will be measured by respiratory indirect calorimetry (Cosmed).
Total energy expenditure | About 14 days.
  Total energy expenditure in kcal or MJ will be measured using the DLW method. TEE will then be calculated using mean CO2 production using the Weir equation.
Environmental temperature | About 14 days.
  The iButton (DS1921G) monitors will be provided for the assessment of both indoor and outdoor temperature of their living environment, measured in degrees Celsius (°C).
Physical activity | About 14 days.
  Physical activity of the participants will be recorded using a GT3X accelerometer worn at the waist for a consecutive period of 14 days. Outcomes measured by the GT3X included physical activity energy expenditure in kcal or MJ, Total MVPA in minutes per day , and Vector Magnitude Counts expressed as counts per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Institutes of Advanced Technology，Chinese Academy of Sciences, Shenzhen, Guangdonng, China

REFERENCES:
- [Background] Speakman JR, Yamada Y, Sagayama H, Berman ESF, Ainslie PN, Andersen LF, Anderson LJ, Arab L, Baddou I, Bedu-Addo K, Blaak EE, Blanc S, Bonomi AG, Bouten CVC, Bovet P, Buchowski MS, Butte NF, Camps SGJA, Close GL, Cooper JA, Creasy SA, Das SK, Cooper R, Dugas LR, Ebbeling CB, Ekelund U, Entringer S, Forrester T, Fudge BW, Goris AH, Gurven M, Hambly C, El Hamdouchi A, Hoos MB, Hu S, Joonas N, Joosen AM, Katzmarzyk P, Kempen KP, Kimura M, Kraus WE, Kushner RF, Lambert EV, Leonard WR, Lessan N, Ludwig DS, Martin CK, Medin AC, Meijer EP, Morehen JC, Morton JP, Neuhouser ML, Nicklas TA, Ojiambo RM, Pietilainen KH, Pitsiladis YP, Plange-Rhule J, Plasqui G, Prentice RL, Rabinovich RA, Racette SB, Raichlen DA, Ravussin E, Reynolds RM, Roberts SB, Schuit AJ, Sjodin AM, Stice E, Urlacher SS, Valenti G, Van Etten LM, Van Mil EA, Wells JCK, Wilson G, Wood BM, Yanovski J, Yoshida T, Zhang X, Murphy-Alford AJ, Loechl CU, Melanson EL, Luke AH, Pontzer H, Rood J, Schoeller DA, Westerterp KR, Wong WW; IAEA DLW database group. A standard calculation methodology for human doubly labeled water studies. Cell Rep Med. 2021 Feb 16;2(2):100203. doi: 10.1016/j.xcrm.2021.100203. eCollection 2021 Feb 16. PMID 33665639
- [Background] WEIR JB. New methods for calculating metabolic rate with special reference to protein metabolism. J Physiol. 1949 Aug;109(1-2):1-9. doi: 10.1113/jphysiol.1949.sp004363. No abstract available. PMID 15394301